CLINICAL TRIAL: NCT01113073
Title: The Distribution of Pressure in the Thorax During Mechanical Ventilation and Its Effects on the Circulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: P. Pickkers MD, PhD, Radboud University Nijmegen Medical Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UMCN_IC_BL_01/2010
Record Dates: First submitted 2010-04-22; First posted 2010-04-29 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-01

CONDITIONS: Fluid Responsiveness
Keywords: pulse pressure variation; hemodynamic monitoring; fluid responsiveness; mechanical ventilation; fluid therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Elective open heart surgery (Experimental): Patients who had undergone elective open heart surgery
  Interventions: Other: ventilatory protocol; Other: Elastic band; Other: passive leg raising test

INTERVENTIONS:
Other: ventilatory protocol — Ventilatory protocol for short period with four different tidal volumes (12 min)
Other: Elastic band — Placement of an elastic band around thorax to reduce thorax compliance
Other: passive leg raising test — performing the passive leg raising test

SUMMARY:
Fluid administration is a daily intervention on the intensive care unit to improve cardiac output (CO) and stabilize circulation in critically ill patients. Simultaneously, the volume status of the patient is very difficult to assess. Too little volume leads to inadequate organ perfusion followed by ischemia and organ failure. Too much volume may worsen heart failure and cause pulmonary and peripheral edema and contribute to further tissue injury and organ dysfunction. Although dynamic indices have been shown to be more accurate predictors of fluid responsiveness, this relevant and complex task is usually guided by static clinical variables and the specialist's interpretation due to the fact that the interpretation of dynamic parameters is not fully developed and that they are not universally available. This lack of understanding is partially because of the complex interaction with mechanical ventilation. The investigators hypothesize that knowing the distribution of ventilatory pressures will make it possible to index dynamic parameters to tidal volume and improve their predictive value concerning the volume status of the patient. In addition, it would be of interest to be able to predict fluid responsiveness in a non-invasive way, especially in critically ill patients. Up to now, continuous non-invasive cardiac output monitoring using Nexfin in critically ill patients has not been validated and also not tested for its ability to predict fluid responsiveness. The present research proposal evaluates the possibility and accuracy of the model flow analysis obtained by non-invasive finger arterial pressure measurements to determine fluid responsiveness using passive leg raising. It will also be compared to a more invasive method (that is currently used in the clinic) to assess its ability to measure absolute CO levels accurately. It may make it possible to assess fluid responsiveness in a non-invasive and patient friendly way.

ELIGIBILITY:
Inclusion Criteria:

* Elective open heart surgery.

Exclusion Criteria:

* Significant cardiac arrhythmias, including atrial fibrillation.
* Hemodynamical instability, as defined by a variation in heart rate, blood pressure and cardiac output of more than 10% during the 15-min period before starting the protocol.
* Recent myocardial infarction (< 3 mnd, troponine > 50 ug/l).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
fluid responsiveness | 30 minutes around fluid challenge
  pulse pressure variation (PPV), systolic pressure variation (SPV), stroke volume variation (SVV), pre-ejection period variation (dPEP)

SECONDARY OUTCOMES:
Pressure distribution in thorax due to mechanical ventilation | 30 minutes of varying tidal volumes
  mechanical ventilation with 4 different tidal volumes and decreased chest compliance
Dynamic indices in pressure support ventilation | 30 minutes of pressure support
non invasive prediction of fluid responsiveness | 30 minutes around fluid challenge
  pulse contour analysis of cardiac output with finger cuff combined with passive leg raising test
pressure distribution and dynamic indices during spontaneous breathing | 5 minutes of spontaneous breathing

CONTACTS AND LOCATIONS:
Overall Officials: Benno Lansdorp, MSc., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands